CLINICAL TRIAL: NCT02735005
Title: Epidemiology of Aging of People With Disabilities - Gerontological Sector "Rumilly-Annecy-Saint-Julien-Pays de Gex-Bellegarde" : Description of the Population in an Attempt to Identify Ways to Implement to Meet the Needs in Aging
Brief Title: Determining the Needs of Aging People With Disabilities
Acronym: PHV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: Agence Régionale de Santé Rhône-Alpes (Other); Conseil Départemental de haute-Savoie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-A00642-47
Record Dates: First submitted 2016-03-24; First posted 2016-04-12 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2018-04

CONDITIONS: Disabled People; Aging; Mental Handicap

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SMAF assessment (Experimental): Face to face interview for the Functional Autonomy Measurement System (SMAF) tool questionnaire For disabled patients living at home, the Social SMAF questionnaire is used in addition.
  Data related to care consumption of each enrolled patients are collected too.
  Interventions: Other: SMAF assessment

INTERVENTIONS:
Other: SMAF assessment — After written information and non opposition expression, each enrolled patient will be assessed with the Functional Autonomy Measurement System (SMAF) tool during a 1 hour interview.
  The French authority has considered this study as an interventional study with minimal risk because we use a tool (SMAF) that was not developped nor validated in this specific population (disabled people older than 40y). The SMAF assessment is not made in routine in this specific population (ID RCB : 2015-A00642-47)

SUMMARY:
Heterogeneous modalities of aging lead to describe three categories of elderly patients: 1-healthy without frailty, 2- healthy with frailty, 3- patients with chronic disease(s) and frailty. Frail people have a high risk of losing functional independence and as a consequence they require more help for day to day life. It is known in elderly that physical activities, nutrition, social environment are important to maintain functional independence.

For patients with disabilities, less is known about the occurence of dependance with aging. That is of growing importance because life expectancy of disabled patients has increased a lot during last decades, and because caregivers, often parents, also become elderly and frail.

So the investigators will require tools to anticipate prevention and supportive needs for this specific population.

The goal of this study is to evaluate if the participants (disabled patients over 40 years old) of a well-defined region in the south-east of France (400000 inhabitants), and to assess their needs, using the Functional Autonomy Measurement System (SMAF) developed for assessment of the elderly, by Rejean Hebert & Nicole Dubuc's team in Sherbrooke University (Quebec/Canada).

ELIGIBILITY:
Inclusion Criteria:

* adult 40 years or older
* must need help allocated by government social health services (Committee on Rights and Autonomy of Disabled People = french CDAPH)
* must live

  1. either in dedicated units or specialized homes (french medicalized care homes, or dedicated community homes)
  2. or at home but working in specialized dedicated centers (So called french Etablissement et Service d'Aide par le Travail) or requiring intervention of specialized services (Support Service for Social Life or Medical-Social Support Service for Disabled Adults)

     Exclusion Criteria:
* patient or patient's legal guardian opposed to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09-26 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Needs in supports for aging disabled patients | through study completion, an average of 1 year
  classification into one of the fourteen homogenous profiles of the Fonctional Autonomy Measurement System (SMAF) tool. The SMAF tool is a software based on responses of 29 predefined items on incapacities (with 4 modalities of response for each) and care and ressources used by interviewed people. The social SMAF tool adds 6 supplementary items (also with 4 modalities of response for each).
  Predefined algorithms defined for not disabled elderly people leads to classification into 14 homogeneous profiles. Progression's modalities of elderly from one profile to another is well known.
  The goal of this study is to determine if the same tool could be used for a younger disabled population, and if not, we want to build other algorithms dedicated to this aging disabled population. That's why this study is performed in collaboration with the Sherbrooke's team who designed the SMAF tool.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu DEBRAY, MD, Principal Investigator — CH Annecy Genevois, head of the gerontological sector; Max BUCHNER, Principal Investigator — Foyer le pré vert - Villeurbanne
Locations (30):
- France (30):
  - FAM du Moulin, Allinges
  - APF - SAVS Annecy, Annecy
  - ESAT "Ateliers de Novel", Annecy
  - FAM Le Goëland, Annecy
  - SAVS - Association Départementale des Infirmes Moteurs Cérébraux, Annecy
  - Savs Archim'Aide, Annecy
  - Savs Espoir 74-Oxygene, Annecy
  - ESAT Bellegarde Industries, Bellegarde
  - EHPAD Maison de Famille du Genevois, Collonges-sous-Salève
  - ESAT Ferme de Chosal, Copponex
  - ADMR Haute-Savoie - SSIAD/SAD, Cran-Gevrier
  - ADTP Site de Cran-Gevrier (Entreprises Adaptées), Cran-Gevrier
  - Esat Messidor, Cran-Gevrier
  - ESAT Antenne du pays de Gex, Ferney-Voltaire
  - Foyer des Roseaux and FAM des Iris, La Balme-de-Sillingy
  - EHPAD La Bartavelle, Meythet
  - FAM Le Goëland, Meythet
  - FAM Résidence Leirens - Armée du Salut Monnetier Mornex, Monnetier
  - SAVS Association Vivre en Ville 01, Ornex
  - ESAT L'Arcalod, Rumilly
  - Association ECLAT Pays de Gex, Saint-Genis
  - FAM Pré la Tour, Saint-Jean
  - ESAT Le Central, Seynod
  - ESAT Le Semnoz, Seynod
  - SAMSAH Le Fil d'Ariane, Seynod
  - SAMSAH Le Bilboquet, Seynod
  - Centre Arthur Lavy - FAM Le Cristal, Thorens-Glières
  - Centre Arthur Lavy - MAS l'Opaline, Thorens-Glières
  - ESAT Myriade, Thônes
  - Association "Nous aussi" - Foyer d'hébergement - SATTHAV, Vétraz-Monthoux

REFERENCES:
- [Background] Ahmed N, Mandel R, Fain MJ. Frailty: an emerging geriatric syndrome. Am J Med. 2007 Sep;120(9):748-53. doi: 10.1016/j.amjmed.2006.10.018. PMID 17765039
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Rubenstein LZ, Josephson KR, Wieland GD, English PA, Sayre JA, Kane RL. Effectiveness of a geriatric evaluation unit. A randomized clinical trial. N Engl J Med. 1984 Dec 27;311(26):1664-70. doi: 10.1056/NEJM198412273112604. PMID 6390207
- [Background] Stuck AE, Siu AL, Wieland GD, Adams J, Rubenstein LZ. Comprehensive geriatric assessment: a meta-analysis of controlled trials. Lancet. 1993 Oct 23;342(8878):1032-6. doi: 10.1016/0140-6736(93)92884-v. PMID 8105269
- [Background] Stuck AE, Egger M, Hammer A, Minder CE, Beck JC. Home visits to prevent nursing home admission and functional decline in elderly people: systematic review and meta-regression analysis. JAMA. 2002 Feb 27;287(8):1022-8. doi: 10.1001/jama.287.8.1022. PMID 11866651
- [Background] Carlsen WR, Galluzzi KE, Forman LF, Cavalieri TA. Comprehensive geriatric assessment: applications for community-residing, elderly people with mental retardation/developmental disabilities. Ment Retard. 1994 Oct;32(5):334-40. PMID 7984118
- [Background] Pinsonnault E, Dubuc N, Desrosiers J, Delli-Colli N, Hebert R. Validation study of a social functioning scale: The social-SMAF (social-Functional Autonomy Measurement System). Arch Gerontol Geriatr. 2009 Jan-Feb;48(1):40-4. doi: 10.1016/j.archger.2007.10.001. Epub 2007 Dec 3. PMID 18061289
- [Background] Dubuc N, Hebert R, Desrosiers J, Buteau M, Trottier L. Disability-based classification system for older people in integrated long-term care services: the Iso-SMAF profiles. Arch Gerontol Geriatr. 2006 Mar-Apr;42(2):191-206. doi: 10.1016/j.archger.2005.07.001. Epub 2005 Aug 25. PMID 16125809
- [Background] Gervais P, Hebert R, Lamontagne J, Tousignant M. [Implementation of functional autonomy measurement system: barriers and facilitators in PISE-Dordogne project]. Geriatr Psychol Neuropsychiatr Vieil. 2011 Dec;9(4):417-28. doi: 10.1684/pnv.2011.0306. French. PMID 22182818
- [Background] Vellas BJ, Wayne SJ, Romero L, Baumgartner RN, Rubenstein LZ, Garry PJ. One-leg balance is an important predictor of injurious falls in older persons. J Am Geriatr Soc. 1997 Jun;45(6):735-8. doi: 10.1111/j.1532-5415.1997.tb01479.x. PMID 9180669
- See also: Loones A, David-Alberola E, Jauneau P (dec 2008). La fragilité des personnes âgées : perceptions et mesures. Centre de Recherche pour l'Étude et l'Observation des Conditions de Vie. Cahier de recherche n°C256 — http://www.credoc.fr/publications/abstract.php?ref=C256
- See also: Pillard F, Rivière D (june 2009). Pratique d'une activité physique ou sportive chez les seniors. Dossier " Activités physiques ou sportives & santé " adsp n° 67 — http://www.hcsp.fr/explore.cgi/Adsp?clef=107
- See also: Haveman M et al 2009 Report on the State of Science on Health Risks and Ageing in People with Intellectual Disabilities.Special Interest Research Group on Ageing and Intellectual Disabilities/Faculty Rehabilitation Sciences University of Dortmund — https://www.google.fr/search?q=Haveman+MJ+et+al+2009+Report+on+the+State+of+Science+on+Health+Risks+and+Ageing+in+People+with+Intellectual+Disabilities.+IASSID+Special+Interest+Research+Group+on+Ageing+and+Intellectual+Disabilities/Faculty+Rehabilitation+Sciences+University+of+Dortmund&ie=utf-8&oe=utf-8&gws_rd=cr&ei=cenyVrC1O4j1aIWQlcAJ
- See also: Rapport Jacob (2013). Un droit citoyen pour la personne handicapée. Un parcours de soins et de santé sans rupture d'accompagnement. — http://www.sante.gouv.fr/IMG/pdf/rapport-pjacob-0306-macarlotti.pdf
- See also: Seematter-Bagnoud L et al (2012). Le Resident Assessment Instrument et autres instruments d'évaluation des personnes âgées. Lausanne : Institut universitaire de médecine sociale et préventive. (Raisons de santé, 191) — http://www.iumsp.ch/Publications/pdf/rds191_fr.pdf
- See also: Gohet P (Nov 2013) L'avancée en âge des personnes handicapées, contribution à la réflexion. — http://social-sante.gouv.fr/ministere/documentation-et-publications-officielles/rapports/handicap/article/l-avancee-en-age-des-personnes-handicapees-contribution-a-la-reflexion